CLINICAL TRIAL: NCT01661010
Title: The Clinical Study of Patients With Sex Chromosome Variants
Brief Title: The Clinical Study of Sex Chromosome Variants
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 120181; 12-HG-0181
Record Dates: First submitted 2012-08-07; First posted 2012-08-09 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2025-08-20

CONDITIONS: Male Factor Infertility; Female Factor Infertility
Keywords: Infertility; Turner Syndrome; X-Chromosome; Y-Chromosome; Aneuploidy; Natural History
MeSH Terms: conditions — Infertility; Turner Syndrome; Aneuploidy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Family members can serve as control group
- Sex-linked genes: Patients previously identified through outside research or diagnostic labs as having sex-chromosome variants causing deletion/duplication of sex-linked genes or entire sex chromosomes.

SUMMARY:
Purpose/Lay Summary: Background:

- Chromosomes are the structures inside of each cell that carry our genetic material (genes). Certain differences in the sex chromosomes are known to cause various diseases, such as infertility, Turner syndrome, or Klinefelter syndrome. However, it is not fully understood why these differences are seen and what clinical findings may be caused with different sex chromosome variants. This study is seeking to learn more about the genetic and clinical characteristics of disorders related to the X and Y chromosomes.

Objectives:

- To study related medical conditions in people with sex chromosome variants.

Eligibility:

* Patients with known sex chromosome differences may be eligible to participate.
* Healthy volunteers age 18 - 55

Design:

* Participants will be screened with a physical exam and medical history. Blood and urine samples will be collected.
* This study will last about 5 days. Participants will have a variety of endocrine and other tests. They will provide blood, urine, and semen samples for these tests.
* Imaging studies of the heart and abdomen will be performed. These tests may include ultrasounds and magnetic resonance imaging.
* Participants will also have their vision and hearing checked.
* Healthy volunteers with have a single day visit for a medical history, physical exam, and blood and skin samples.
* Treatment will not be provided as part of this study.
* Compensation is offered.

DETAILED DESCRIPTION:
Infertility is a disease that affects approximately 10% of couples world-wide. Causes of infertility are varied and include age-related decline in fecundity, other causes of ovulatory dysfunction, tubal and pelvic pathology, male causes, idiopathic, and multifactorial. The underlying genetic causes of infertility are incompletely understood. The purpose of this study is to increase our understanding of the genetic and clinical manifestations of infertility related to sex-chromosome variants through detailed physical, radiologic, and laboratory studies. We will concentrate on a group of patients (both male and female) with known sex-chromosome variationsfully characterized through genetic sequencing and karyotyping. Other patients with

sex chromosome variants will be invited depending on the variant described. Patients recruited and consenting to this study will be evaluated at the NIH Clinical Center

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Patients previously identified through outside research or diagnostic labs as having sex-chromosome variants causing deletion/duplication of sex-linked genes or entire sex chromosomes, male and female.
  2. In the event that a patient with a sex-chromosome variant self-refers to the protocol, medical records will be reviewed by a committee to include Dr. David Page, Dr. Maximilian Muenke, and others to decide whether the patient is appropriate for enrollment in the protocol.
  3. Willing family members of subjects enrolled may be enrolled as control subjects.

EXCLUSION CRITERIA:

1. We reserve the right to exclude patients with medical conditions that would place a potential participant at high risk of complications if managed at the NIH clinical center (ex. dialysis dependency, unstable cardiac conditions, unstable severe depression/suicidality).
2. We reserve the right to exclude cases that are clearly not related to sex-chromosome variants, infertility or our direct research interests (e.g. infertility with clearly non-genetic etiology). This almost never happens, and we would attempt to make referrals to a more

appropriate investigator.

It is our intention to try to remove as many economic, cultural, geographic, racial, and gender barriers as we reasonably can to promote a diverse participation of sex-chromosome variant cases for research purposes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients previously identified through outside research or diagnostic labs as having sex-chromosome variants causing deletion/duplication of sex-linked genes or entire sex chromosomes.@@@
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2012-07-30 (Actual)

PRIMARY OUTCOMES:
Phenotype | Ongoing
  To characterize the physical, reproductive, endocrinologic and radiologic phenotype of a group of patients who have known sex-chromosome structural and copy-number variants.
Spectrum | Ongoing
  To examine the spectrum of clinical characteristics of infertility and other conditions related to sex-chromosome variants and facilitate early clinical recognition, diagnostic confirmation, anticipatory management, prognostication, and proper genetic counseling.

CONTACTS AND LOCATIONS:
Overall Officials: Ashley J Buscetta, C.R.N.P., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Brandell RA, Mielnik A, Liotta D, Ye Z, Veeck LL, Palermo GD, Schlegel PN. AZFb deletions predict the absence of spermatozoa with testicular sperm extraction: preliminary report of a prognostic genetic test. Hum Reprod. 1998 Oct;13(1O):2812-5. doi: 10.1093/humrep/13.10.2812. PMID 9804236
- [Background] Bondy CA; Turner Syndrome Study Group. Care of girls and women with Turner syndrome: a guideline of the Turner Syndrome Study Group. J Clin Endocrinol Metab. 2007 Jan;92(1):10-25. doi: 10.1210/jc.2006-1374. Epub 2006 Oct 17. PMID 17047017
- [Background] Berta P, Hawkins JR, Sinclair AH, Taylor A, Griffiths BL, Goodfellow PN, Fellous M. Genetic evidence equating SRY and the testis-determining factor. Nature. 1990 Nov 29;348(6300):448-50. doi: 10.1038/348448A0. PMID 2247149
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-HG-0181.html